CLINICAL TRIAL: NCT01594034
Title: Effects of Hemoperitoneum Driven Carbon Monoxide on Post-Traumatic Stability
Brief Title: Effects of Hemoperitoneum Driven Carbon Monoxide on Post-Traumatic Stability and Platelet Aggregation
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-2009-0176-H
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Hemoperitoneum
MeSH Terms: conditions — Hemoperitoneum

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment
  Interventions: Procedure: expired air

INTERVENTIONS:
Procedure: expired air — collection of expired air from ventilator

SUMMARY:
Our objective is to determine whether or not the presence of hemoperitoneum in trauma patients is associated with increased Carbon Monoxide (CO) formation, and to determine if elevated Carbon Monoxide levels are associated with cardiovascular depression, impaired platelet aggregation, and/or multiple organ failure.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized males 18 years of age or older,
2. Diagnosis of isolated blunt OR blunt and penetrating trauma,
3. Admitted or expecting to be admitted to the Intensive Care Unit,
4. On mechanical ventilation, and
5. Written informed consent obtained

Exclusion Criteria:

1. Female gender, (Females will be excluded from this study as the menstrual cycle and other estrogen variations are known to be associated with cyclic changes in CO production adding a potential confounder to the interpretations of our findings.)
2. Diagnosis of isolated penetrating trauma,
3. Acute hemothorax or pneumothorax,
4. Treatment with antiaggregants (ASA, clopidogrel, aggrenox or ticlopidine),
5. Enrollment in another research study,
6. Prisoners,
7. Inability to perform CO measurement within 96 hours after hospital admission.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in the ICU on a ventilator
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
•Establish a method for reliably measuring CO excretion in patients. | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Johnson, PhD, Principal Investigator — University of Texas
Locations (1):
- University Hospital, San Antonio, Texas, United States